CLINICAL TRIAL: NCT07256808
Title: Efficacy of a Lower Leg Strengthening Program in the Prevention of MTSS in Collegiate XC Runners
Brief Title: Medial Tibial Stress Syndrome Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rowan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro-2023-75
Record Dates: First submitted 2025-05-11; First posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-05

CONDITIONS: Medial Tibial Stress Syndrome
MeSH Terms: conditions — Medial Tibial Stress Syndrome | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resistance Training Intervention (Experimental): Participants who received the heavy resistance training intervention in addition to their regular training.
  Interventions: Other: Resistance Training
- Regular Training (No Intervention): Participants who continued their regular training without the additional intervention.

INTERVENTIONS:
Other: Resistance Training — Participants performed a 10-week resistance training program, completing exercises twice daily for Weeks 1-2 and three times daily for Weeks 3-10, with 5 sessions per week for Weeks 1-7 and 6 sessions per week for Weeks 8-10. The program included exercises such as standing broad jumps, resisted ankle abduction, single-leg eccentric plantar flexion, and ankle rockers. Participants' muscle properties were assessed at the start and end of the intervention, with adherence monitored via remote video confirmation.
  Arms: Resistance Training Intervention

SUMMARY:
This randomized controlled trial investigated whether a 10-week heavy resistance training program reduced the incidence of medial tibial stress syndrome (MTSS) in collegiate indoor track and field athletes. Twenty-six athletes from Rowan University were randomly assigned to a treatment group (resistance training plus regular training) or a control group (regular training only). Muscle mechanical properties-including tone, stiffness, elasticity, stress relaxation time, and creep-were measured by MyotonPro device (non-invasive) at baseline, post-intervention, and at the end of the season. A 10-week observational follow-up during the indoor season included weekly MTSS symptom surveys. Differences in MTSS incidence and muscle properties were analyzed between groups.

ELIGIBILITY:
Inclusion Criteria:

* Collegiate athletes on the Indoor Track and Field team.
* Athletes must participate in at least one of the following:
* 60m-800m events (including hurdles)
* jumping events (including pole vault)

Exclusion Criteria:

* Subjects who have a history of musculoskeletal or neurologic conditions
* Who take medications that affect muscle tone
* Who have a body mass index >30.0 kg/m2 were excluded to screen to prevent adipose tissue from skewing the measurements.
* Any subject with any fractures, sprains, or strains of the lower extremities were excluded.
* Any subject with active MTSS, stress fracture, or other lower leg pathology symptoms at the time the initial survey was administered were excluded.
* Any athlete who does not participate in the 60m-800m events (including hurdles), or who does not participate in jumping events (including pole vault) were excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2023-09-14 (Actual); Primary Completion 2024-02-14 (Actual); Study Completion 2024-02-14 (Actual)

PRIMARY OUTCOMES:
Subjective Medial Tibial Stress Syndrome Symptoms | Through the running season -- approximately 11 weeks
  Medial Tibial Stress Syndrome (MTSS) Score Survey

SECONDARY OUTCOMES:
Myotonometry Oscillation frequency | From enrollment through the end of data collection -- approximately 25 weeks
  Represents the intrinsic tension of the muscle in its passive state, essentially the muscle's "tone".
Myotonometry dynamic stiffness | From enrollment through the end of data collection -- approximately 25 weeks
  Measures the resistance of the tissue to deformation when subjected to an external force.
Myotonometry logarithmic decrement | From enrollment through the end of data collection -- approximately 25 weeks
  Indicates the elasticity of the muscle
Myotonometry mechanical stress relaxation time | From enrollment through the end of data collection -- approximately 25 weeks
  Measures the time it takes for the muscle to return to its original shape after being deformed.
Myotonometry creep | From enrollment through the end of data collection -- approximately 25 weeks
  Describes the gradual elongation of the muscle under constant tensile stress over time.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer A Longo, PhD, Principal Investigator — Rowan University
Locations (1):
- Rowan University, Glassboro, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No